CLINICAL TRIAL: NCT06686953
Title: Clinical Study of the Effect of Environmental Pollution on the Prognosis of Colorectal Cancer.
Brief Title: The Effect of Environmental Pollution on Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: ZZ2024-291-01
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Carcinoma
Keywords: colorectal cancer; environment; airpollution; greenness
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- the colorectal cancer group: patients diagnosed as colorectal cancer

SUMMARY:
Colorectal cancer (CRC) is one of the most common malignancies worldwide, and its main risk factors include age, genetic factors, inflammatory bowel diseases (e.g., ulcerative colitis and Crohn's disease), unhealthy diets (e.g., high-fat, low-fibre diets), obesity, physical inactivity, smoking, and excessive alcohol consumption. The relationship between environmental pollution and colorectal cancer has received increasing attention in recent years. Studies have shown that long-term exposure to fine particulate matter in the air, such as passive smoking, soot and oil smoke exposure, incense burning exposure, occupational exposure and outdoor work, PM2.5, PM10 and NO2 may increase the risk of colorectal cancer. These particulate matter can enter the lungs through breathing and trigger a chronic inflammatory response in the systemic system, thus increasing the risk of cancer development. This study intends to determine the extent of air pollution's impact on colorectal cancer prognosis by analysing survival data of colorectal cancer patients in regions with different pollution levels. As well as to investigate the association between air pollution levels and postoperative recurrence in colorectal cancer patients, looking for possible mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* patients diagnosed with colorectal cancer by pathological biopsy before surgery;
* patients did not undergo chemotherapy, radiotherapy, targeted and immunotherapy, etc. before enrolment;
* willing to participate in this study and sign an informed consent form;
* complete clinical data.

Exclusion Criteria:

* patients with primary malignant tumours other than colorectal cancer;
* patients with systemic diseases, such as severe cardiopulmonary insufficiency, that affect the choice of treatment options;
* patients who are not suitable for enrolment as assessed by the investigator;
* incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed as colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 6300 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
colorectal cancer | From 18 years old until the developing colorectal cancer, through study completion, an average of 5 year.
  the time for diagnosing colorectal cancer

IPD SHARING:
Plan to Share IPD: No
Clinical centres conducting this study are not allowed to disclose patient information and data sharing.